CLINICAL TRIAL: NCT05264974
Title: Novel RNA-lipid Particle (RNA-LP) Vaccine for Anti-PD-1 Antibody Therapy Sensitization
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UF-CUT-001; IRB202200462 (Other: University of Florida); OCR41806 (Other: University of Florida)
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Melanoma; Soft Tissue Sarcoma
Keywords: melanoma; immunotherapy; vaccines; RNA-NP; soft tissue sarcoma
MeSH Terms: conditions — Melanoma; Sarcoma | interventions — Nanoparticles; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mRNA-nanoparticle (mRNA-NP) vaccine (Experimental)
  Interventions: Biological: Autologous total tumor mRNA loaded DOTAP liposome vaccine

INTERVENTIONS:
Biological: Autologous total tumor mRNA loaded DOTAP liposome vaccine — All participants will receive three doses of RNA-NP vaccine (1 dose every 2 weeks) intravenously.
  The vaccine dose given will be determined by a 3 + 3 design. Participants will be given one of the following vaccine doses:
  Dose level 0 (starting dose level): 0.00125 mg/kg mRNA in 0.01875 mg/kg LP; Dose level 1: 0.0025 mg/kg mRNA in 0.0375 mg/kg LP; Dose level 2: 0.005 mg/kg mRNA in 0.075 mg/kg LP; or Dose level 3: 0.01 mg/kg mRNA in 0.15 mg/kg LP
  If 3 or more of the initial 6 subjects experience a dose-limiting toxicity, then the initial starting dose will be reduced (dose de-escalation) to 0.000625 mg/kg mRNA encapsulated in 0.009375mg/kg LPs (Dose level -1).
  Other Names: mRNA-NP (nanoparticle) vaccine

SUMMARY:
The goal of this phase I trial is to evaluate the toxicity and feasibility of a tumor-specific RNA-NP vaccine in patients with stage IIB-IV melanoma who have evidence of progressive disease by RECIST 1.1 criteria while receiving adjuvant aPD1 therapy, or those who progress within 6 months of completion of adjuvant treatment, or unresectable stage II soft tissue sarcoma or stage III-IV soft tissue sarcoma.

DETAILED DESCRIPTION:
Melanoma is an increasing public health concern in the state of Florida. The advent of immune checkpoint inhibitors (ICI) has revolutionized the treatment of advanced melanoma. Unfortunately, in the adjuvant setting, up to 30% of subjects will have disease recurrence within 1 year of starting ICI therapy. Previous studies have shown that subjects who progress while on adjuvant ICI treatment, or soon after completion, have a more aggressive course of disease that responds poorly to subsequent immunotherapy. One reason for the failure of ICI in the post adjuvant setting is the immune suppressive nature of the tumor microenvironment (TME) and lack of professional APC activation. These APCs remain in an inert state unable to present tumor antigens for immune detection due to lack of innate immune activation and inhibition from myeloid derived suppressor cells (MDSCs). Similarly, outside of rare subtypes, soft tissue sarcomas (STS) are enriched with an immunosuppressive TME leading to resistance to ICI therapy.

We have developed a novel RNA-lipid particle (RNA-LP) vaccine that simultaneously penetrates and reprograms the TME while inducing a tumor specific adaptive T cell response. This vaccine utilizes novel engineering design that layers tumor derived mRNA into a lipid-nanoparticle "onion-like" package along with pp65 full length lysosomal associated membrane protein (LAMP1) mRNA. These RNA-LPs localize to the TME and activate multiple innate pathways thereby activating APCs and suppressing the function of MDSCs. LAMP mRNA is added to improve innate activation as seen in preclinical modeling and to allow for tracking of T cell receptor specific immune response to vaccination. In this study we propose the use of subject derived RNA-LP vaccine in subjects who progress on, or soon after completion of adjuvant ICI. We propose that through re-priming of the antitumor immune response and alteration of the TME we can improve the efficacy of ICI therapy.

If effective, this treatment will revolutionize the management of this aggressive subset of melanoma and STS to improve overall survival. This study will also gather important information into the mechanisms of early ICI resistance, identify novel biomarkers of innate cell resistance and response to treatment, and provides a cutting edge, personalized immunology approach to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old
* ECOG performance ≤ 2
* Lab values within the specified ranges:

  * Hemoglobin ≥ 8G/DL
  * Platelets ≥ 150 thou/cumm
  * Absolute Neutrophil Count (ANC) ≥ 1500 thou/cumm
  * Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * AST and ALT ≤ 2.5 x ULN; If confirmed liver metastases: AST and ALT ≤ 5 x ULN
  * Creatinine clearance (CrCl) ≥ 15 ml/min (based on modified Cockcroft and Gault formula)
* Must have disease that is amenable to surgical sampling for RNA extraction, amplification, and loading of lipid particles
* Subjects must not have more than one active malignancy at the time of enrollment (subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician and approved by the PI] may be included)
* Written informed consent obtained from the subject.
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening
* Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least four months after the last dose of study treatment to minimize the risk of pregnancy. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for four months following the last dose of study treatment and must agree to not donate sperm during the study treatment period or for four months following the last dose of study treatment.

Additional eligibility criteria for subjects with melanoma:

* Must have measurable disease with evidence of progression (progressive disease, or PD) by RECIST 1.1 criteria while receiving adjuvant aPD1 therapy, or progression within 6 months after completing adjuvant treatment for stage IIB-IV melanoma
* Patients with stage IV nonresectable disease with rare melanoma subtypes: (mucosal, acral, uveal, non-sun exposed) are eligible for the study if they fail to response to initial immunotherapy given in the first line metastatic setting. These rare subtypes do not respond to aPD1 blockade at the same rate or degree as cutaneous melanomas and behave more like adjuvant failure patients in response to aPD1. These patients must have disease amenable to sampling and in the opinion of the treating physician have appropriate bridging therapy available to reach vaccination series, have no other approved therapeutic options/or decline their use.
* Patients of any stage treated with immune checkpoint inhibition with primary or secondary immunotherapy resistance. Primary resistance is defined as a minimum drug exposure requirement of 8-12 weeks or roughly two doses of the immunotherapy with Lack of benefit defined as progressive disease at the time of the first planned assessment or stable disease lasting less than 6 months. Secondary resistance is defined as exposure to immune checkpoint inhibition for at least 6 months with best response initially including a complete response, partial response, or stable disease lasting for greater than 6 months with subsequent progression while receiving checkpoint inhibition, or within 6 months of completing a planned course of immunotherapy. These patients are eligible for enrollment if their disease is amenable to sampling for vaccine generation and they are not contraindicated to continuation of immune checkpoint therapy, and do not have rapidly progressing disease, and have no other viable clinical options or choose not to pursue current approved salvage options for therapy.
* Must have received either aPD1, combination aPD1/CTLA-4 inhibition, or PD1/LAG-3 inhibitor as adjuvant or definitive metastatic treatment for stage IIB-IV melanoma following surgical resection
* Must be BRAF wildtype, or have BRAF mutation but contra-indication to BRAF/MEK inhibitor use, have progressed while on BRAF/MEK therapy, or decline the option to utilize BRAF/MEK therapy.

Additional eligibility criteria for subjects with soft tissue sarcoma:

* Must have measurable disease and tumor accessible for tissue sampling
* Evidence of spindle cell, pleomorphic, round cell, or epithelioid morphology on pathology suggestive of sarcoma as determined by a sarcoma pathologist
* Original tumor site from soft tissue location i.e. lipomatous tissue, musculature, skin
* Evidence of unresectable stage II disease; stage III or stage IV disease
* Subjects may be eligible without receiving prior therapy if no FDA approved or standard of care therapy is indicated/available
* Subjects with prior immune checkpoint inhibitor exposure may be eligible, but prior exposure is not required unless it is a component of an FDA approved indication

Exclusion Criteria:

* Subjects that have an active second malignancy, however, previously treated early stage malignancies with no evidence of disease recurrence after 3 years of follow-up will be allowed
* Subjects with a history of immune-mediated treatment-related adverse reactions leading to discontinuation of prior aPD1 therapy or severe hypersensitivity reaction to any monoclonal antibody or any other baseline risk in the opinion of the investigator that precludes continued use of aPD1 therapy
* Patients with active and symptomatic brain metastases or leptomeningeal metastases at time of inclusion. Patients with isolated brain lesions that have been treated with stereotactic radiosurgery or surgical resection as part of oligometastatic initial management prior to start of immunotherapy may be eligible as long as they have no new disease and are asymptomatic at time of inclusion.
* If patients develop new brain metastases during the time between tumor sampling and vaccine generation and administration, patients may remain on study as long as they can receive definitive stereotactic radiosurgery or surgery to brain metastases and be able to resume systemic therapy within 6 weeks of discovery of new brain metastases.
* Subjects who received an investigational drug in another clinical trial must wait 28 days or at least 5 half-lives of the study drug, whichever is shorter, prior to enrollment in this study
* Patients must not have required corticosteroids (anything greater than 10mg of prednisone of equivalent, daily) or other immunosuppressive medications within 14 days of the start of trial treatment.
* Subjects with uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within seven days prior to tissue collection for vaccine creation or within seven days prior to vaccine administration (subjects on prophylactic agents are acceptable)
* Subjects with any life-threatening illness, medical condition, or organ system dysfunction, which in the investigator's opinion, could compromise subject safety
* Subjects with known active hepatitis B virus or untreated hepatitis C virus. Patients with previous history of hepatitis C who completed treatment for HCV would not be excluded as long as they have no detectable viral load.
* Clinically relevant active autoimmune disease that would pose significant risk to the patient's life should a flare ensue. Patients with chronic autoimmune rheumatologic endocrine, or psoriatic skin diseases may still be eligible pending they are not receiving systemic immunosuppression at the time of treatment as previously described and that patients are aware of the increased risk of flare provocation with treatment.
* Symptomatic congestive heart failure (NYHA Class 3 or 4)
* Subjects with unstable angina pectoris
* Subjects who are post-splenectomy, otherwise asplenic, or have moderate to severe splenomegaly (defined as a spleen larger than 13 cm in cranial-caudal height or longest diameter)
* Personal history of anaphylactic reaction to previous vaccination
* Known hypersensitivity to the active substance or to any of the excipients
* Subjects with known human immunodeficiency virus with CD4+T cells ≤ 350 cells/ul, a positive viral load as determined by institutional standard testing, or a history of AIDS defining opportunistic infection within the last 12 months
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 months after the last dose of study treatment
* Females who are confirmed to be pregnant or breastfeeding
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician
* Administration of a vaccine containing live virus within 30 days prior to the first dose of trial treatment. Note: Most flu vaccines are killed viruses, with the exception of the intra-nasal vainer (Flu-Mist) which is an attenuated live virus and therefore prohibited for 30 days prior to first dose. Non-live versions of the COVID vaccine are allowed.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects with sarcoma originating from bone or cartilage
* Sarcomatous malignancies lacking metastatic potential i.e. well-differentiated liposarcoma, dermatofibrosarcoma protuberans, desmoid fibromatosis, etc.
* Subjects with sarcoma who have received dual checkpoint inhibition are not eligible

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 2 months
  Determine the maximum tolerated dose of RNA-NP vaccine
Feasibility of treatment with RNA-NP vaccine | 4 weeks
  Determine the feasibility of treatment with RNA-NP vaccine, defined as the percentage of subjects who undergo tumor sampling and vaccine generation who can have sufficient vaccine produced for treatment across the full three dose vaccination series and within a time window of 4 weeks from time of tumor sampling to vaccine delivery for use.

SECONDARY OUTCOMES:
Overall response rate | 4 weeks
  Determine the overall response rate, defined as the percentage of subjects who attain either a complete or partial response by RECIST 1.1 criteria following completion of the three dose vaccination series.
Progression-free survival | 5 years
  Determine the the rate of progression free survival (PFS), defined as the time from study enrollment until progression, following resumption of immune checkpoint inhibition following RNA-LP vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Leighton Elliott, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Villanueva MT. RNA delivery heats up cold tumours. Nat Rev Drug Discov. 2024 Jul;23(7):497. doi: 10.1038/d41573-024-00098-0. No abstract available. PMID 38858569